CLINICAL TRIAL: NCT07153978
Title: Safety of Thulium Fiber Laser Litothripsy in the Management of Large Renal Stones (>1000 mm³) and Factors Affecting Treatment Success:
Brief Title: Safety of Thulium Fiber Laser Litothripsy in the Management of Large Renal Stones (>1000 mm³) and Factors Affecting Treatment Success
Acronym: RIRS and TFL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muharrem Baturu (Other)
Collaborators: University of Gaziantep (Other)
Responsible Party: Sponsor-Investigator, Muharrem Baturu, assistant professor, University of Gaziantep
Organization: University of Gaziantep (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023/06; TF.ALT.23.10 (Other Grant/Funding Number: GAZİANTEP ÜNİVERSİTESİ - BİLİMSEL ARAŞTIRMA PROJELERİ KOORDİNASYON BİRİMİ)
Record Dates: First submitted 2025-07-17; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Renal Stones; Retrograde Intrarenal Surgery; Thulium Fiber Laser
Keywords: Retrograde intrarenal surgery,; Thulium fiber laser; Stone free rate; Kidney stone; Hounsfield Unit.
MeSH Terms: conditions — Nephrolithiasis; Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Safety and Efficacy of Thulium Fiber Laser for Large Renal Stones (Experimental): Demographic data (age, gender, body mass index (BMI)), stone characteristics (size, location, Hounsfield Unit (HU) value) and durations of the procedures were recorded. Patients over 18 years of age, with kidney stones larger than 1000 mm³, single or multiple stones and those eligible for RIRS were included in the study. Patients under 18 years of age, those with bleeding diathesis or inability to discontinue anticoagulant/antiaggregant therapy, cases with a history of previous RIRS, individuals who did not attend follow-up visits, patients in whom postoperative residual stone assessment could not be made, or had concomitant bladder or ureteral stones were excluded. SFRs, the need for a second session of RIRS and complications were noted. General anesthesia was used. Rigid ureteroscope was inserted through urethral meatus. 11/13 F ureteral sheath was advanced over guidewire under fluoroscopy. Laser settings varied 0.2J/100Hz to 1J/10Hz based on stone fragility.
  Interventions: Device: Effectivity of TFL on large renal stone

INTERVENTIONS:
Device: Effectivity of TFL on large renal stone — While literature studies on TFL have focused on the effect of stone size on laser efficacy parameters, the present study is important as it is a prospective study examining the effects of TFL lithotripsy on SFRs in stones >1000 mm3.

SUMMARY:
The aim of this study is to compare the efficacy and safety of Thulium Fiber Laser (TFL) litothripsy according to stone density and the factors affecting success in patients undergoing retrograde intrarenal surgery (RIRS) for renal calculi >1000 mm3. Between November 2023 and December 2024, 81 patients with a stone volume >1000 mm3 who underwent RIRS with TFL in our clinic were prospectively and sequentially evaluated. Stone density of the patients was measured, and expressed in Hounsfield Units (HU). Patients with stone densities <1000 HU and ≥1000 HU were categorized as Groups 1, and 2, respectively. Demographic data, data of intraoperative laser use, stone-free rates (SFRs), the need for a second session of RIRS and complications were recorded. Duration of TFL litothripsy, total energy used, laser ablation speed (mm3/sec), laser ablation efficiency (mm3/J) and laser energy consumption (J/mm3) were calculated. Correlation tests, univariate and multivariate logistic regression tests were used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age
* Presence of kidney stones larger than 1000 mm³
* Patients with single or multiple kidney stones
* Patients eligible for retrograde intrarenal surgery (RIRS)

Exclusion Criteria:

* Patients younger than 18 years
* Pregnant or breastfeeding women
* Patients with uncorrected coagulopathy
* Patients with active urinary tract infection
* Patients with severe anatomic abnormalities preventing RIRS
* Patients unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome was to assess the effectiveness of the laser. | 12 months
  Fragmentation success was used to evaluate the laser effectiveness of laser.

SECONDARY OUTCOMES:
The secondary outcome was the evaluation of factors affecting stone-free rates | 3 months
  A residual fragment of ≤2 mm was considered stone-free. The unit of measure for all parameters was the percentage of patients stone-free.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Gaziantep, Gaziantep, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP